CLINICAL TRIAL: NCT00889421
Title: An Open-label Trial to Assess the Efficacy and Safety of Apremilast in the Management of Vision-threatening Uveitis That is Refractory to Other Modes of Systemic Immunosuppression.
Brief Title: Apremilast in the Treatment of Uveitis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Investigator discretion due to lack of efficacy in three subjects enrolled
Sponsor: Oregon Health and Science University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Eric B. Suhler, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: e4235
Record Dates: First submitted 2009-04-24; First posted 2009-04-28 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Uveitis
Keywords: uveitis; apremilast
MeSH Terms: conditions — Uveitis | interventions — apremilast

ARMS (1):
- Treatment (Experimental): Patients receiving apremilast.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — oral dose of 30 mg BID for 6 months

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Apremilast in the treatment of uveitis.

ELIGIBILITY:
Inclusion Criteria:

* patients with vision-threatening autoimmune uveitis
* failure to respond to prednisone and at least one other systemic immunosuppressive, or intolerance to such medications due to side effects

Exclusion Criteria:

* serious concomitant illness that could interfere with the subject's participation
* previous or current use of an alkylating agent
* use of CYP3A4 inhibitors during the trial
* TNF blocker use within the 8 weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric B Suhler, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Patient receiving apremilast.
Period: Overall Study
Arm/Group | Treatment
Started | 3
Completed | 0
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Population: patients with refractory uveitis
Arm/Group | Treatment
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Improvement by 2 or More Lines of Best-corrected Snellen Visual Acuity in at Least One Eye
Time Frame: 6 months
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Primary Outcome: Reduction in Dose of Systemic Corticosteroid or Other Immunosuppressive Therapy by at Least 50%
Time Frame: 6 months
Arm/Group | Treatment
Number analyzed (Participants) | 0

3. Primary Outcome: Control of Ocular Inflammation, as Judged on Clinical Criteria, According to Standard Methods (Reduction of Anterior Chamber Cellular Activity and/or Chorioretinal Infiltrates and/or Retinal Vasculitis)
Time Frame: 6 months
Arm/Group | Treatment
Number analyzed (Participants) | 0

4. Primary Outcome: Reduction in Cystoid Macular Edema
Time Frame: 6 months
Arm/Group | Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Type, Frequency, Severity, and Relationship of Adverse Events to Study Treatment
Time Frame: 7 months
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=3)
nausea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated prematurely due to inefficacy in the three initial patients enrolled. Endpoints were not analyzed as participants did not make it to the 6 month time frame before discontinuing the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes